CLINICAL TRIAL: NCT01739023
Title: The Safety of Autologous Human Schwann Cells (ahSC) in Subjects With Subacute Spinal Cord Injury (SCI)
Brief Title: Safety of Autologous Human Schwann Cells (ahSC) in Subjects With Subacute SCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: W. Dalton Dietrich (Other)
Collaborators: The Miami Project to Cure Paralysis (Other)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor of Neurosurgery, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20081061
Expanded Access: NCT02480777 (No longer available)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Spinal Cord Injury; Paraplegia
Keywords: paraplegia; cell therapy; Schwann cells; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Human Schwann Cells (Experimental)
  Interventions: Biological: Autologous Human Schwann Cells

INTERVENTIONS:
Biological: Autologous Human Schwann Cells — Schwann cells harvested from the sural nerve of the participant will be autologously transplanted into the epicenter of the participant's spinal cord injury.

SUMMARY:
The purpose of this study is to assess the safety of autologous human Schwann cells (ahSC) transplantation in subjects with subacute SCI.

For humans with subacute SCI, we hypothesize that axons might show improved function if myelin repair is induced with the implantation of ahSC. In addition spinal cord cavitation may be reduced, and neural sprouting and plasticity may be enhanced via neurotrophic effects.

DETAILED DESCRIPTION:
Schwann cells are excellent candidates for transplantation into humans with SCI. Large numbers of ahSC can be derived for autologous implantation after a minor surgery for peripheral nerve harvesting, and purification and expansion of the cells in culture. Autologous cells offer important safety advantages that include no need for immune suppression, minimal risk of disease transfer, and a low risk of tumorigenicity.

Since 1990, scientists at the Miami Project to Cure Paralysis have generated extensive preclinical data suggesting Schwann cell transplantations are successful in rodents with SCI. The most recent work has focused on contusive injury models that are relevant to human injury. They have also been largely responsible for developing an efficient method for procuring large, essentially pure populations of human Schwann cells from adult peripheral nerve.

The rationale for implantation of ahSC in people with acute SCI is based on the evidence that Schwann cells are neuroprotective and are capable of myelinating axons. Using mitogen expanded human Schwann cells in SCID mice and athymic female nude rats demonstrated that human Schwann cells can survive and are capable of enhancing axonal regeneration and forming myelin after transplantation in animals with sciatic nerve transection or thoracic spinal cord transection. The proposed clinical trial will advance knowledge about the safety and feasibility of a cell-based treatment strategy for human SCI.

This Phase 1 clinical trial will employ an open label, unblinded, nonrandomized and non-placebo controlled dose-escalation design to evaluate the safety of transplantation of ahSC transplantation in subjects with subacute SCI.

A sural nerve harvest will occur within 30 days post-injury. Standard-of-care medical treatment and rehabilitation will proceed while the cells are being processed in a cGMP facility. No later than 72 days post-injury, the ahSC product will be administered via a single injection into the cavity of the spinal cord lesion.

Safety and efficacy assessments will be performed at week 1 and 2 post-transplantation and 2, 6, and 12 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Persons with traumatic SCI that occurred within the previous 30 days.
* 2) Between the ages of 18 and 60 at last birthday.
* 3) SCI at a thoracic level between T3-T11 as defined by MRI and the most caudal level of intact motor and sensory function on the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI).
* 4) Acute SCI with ISNCSCI grade A impairment at time of enrollment.

Exclusion Criteria:

* 1) Persons with penetrating injury of the spinal cord or complete transection of the cord, including bone fragment lacerations, as identified by magnetic resonance imaging (MRI).
* 2) Persons with a lesion in the conus medullaris, cauda equina, or lower extremity peripheral nerve.
* 3) Persons unable to safely undergo an MRI.
* 4) Persons in whom adequate MRI imaging cannot be obtained.
* 5) Persons who have developed a pulmonary embolism (PE) or deep vein thrombosis (DVT).
* 6) Other traumatic injuries (e.g., CHI, another level of SCI) affecting the ability to provide informed consent and participate fully in rehabilitation.
* 7) Persons with self-reported persistent severe neuropathic pain, inadequately controlled by non-narcotic medication.
* 8) Persons with severe persistent mechanical or thermal hypersensitivity/allodynia at the neurological level or rostral to it as documented by clinical testing.
* 9) Pregnant women or a positive pregnancy test in those women with reproductive potential prior to enrollment.
* 10) Presence of systemic disease that might interfere with subject safety, compliance, or evaluation of the condition under study.
* 11) Presence of any unstable medical or psychiatric condition that could reasonably be expected to subject the participant to unwarranted risk from participation in the study or result in a significant deterioration of his/her clinical course.
* 12) Body Mass Index (BMI) > 35.
* 13) History of active substance abuse.
* 14) Persons who have participated in other experimental treatments within the past 90 days deemed by the PI to represent a possible confound or enrolled in any other ongoing trial.
* 15) Persons with significant lower extremity injury, previous surgery, or amputation such that would preclude satisfactory sural nerve harvest.
* 16) Persons allergic to gentamicin
* 17) Persons who test positive for HIV or Hepatitis B or C virus.
* 18) Baseline entry criteria for renal function, CBC, INR, and liver tests including serum albumin, total bilirubin, alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphastase (ALP), and gamma glutamyl transpeptidase (GGT). Persons with lab values that are concerning in the context of SCI may be excluded from participating in the trial if these indicate chronic or severe acute pathology.
* 19) Persons with autoimmune diseases, for which chronic corticosteroids or immunosuppression therapy may be needed.
* 20) Persons with clinically documented malignancy in the past 5 years except for treated non-melanoma skin cancers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
International Standards of Neurological Classification for Spinal Cord Injury | Change from Baseline at 12 months
MRI of spinal cord | Change from Baseline at 12 months
Neuropathic pain | Change from Baseline at 12 months

SECONDARY OUTCOMES:
Spinal Cord Independence Measure III | Change from Baseline at 12 months
Functional Independence Measure | Change from Baseline at 12 months
Motor Evoked Potentials | Change from Baseline at 12 months
Somatosensory Evoked Potentials | Change from Baseline at 12 months
Autonomic - Head-up Tilt | Change from Baseline at 12 months
Autonomic - Sympathetic Skin Response | Change from Baseline at 12 months
ISCI Basic Bowel Dataset | Change from Baseline at 12 months
ISCI Basic Lower Urinary Tract Dataset | Change from Baseline at 12 months
SF-12 | Change from Baseline at 12 months
Patient Global Impression of Change | Change from Baseline at 12 months
Modified Ashworth Scale | Change from Baseline at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dalton Dietrich, PhD, Study Director — University of Miami; Allan Levi, MD, PhD, Principal Investigator — University of Miami; James Guest, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Anderson KD, Guest JD, Dietrich WD, Bartlett Bunge M, Curiel R, Dididze M, Green BA, Khan A, Pearse DD, Saraf-Lavi E, Widerstrom-Noga E, Wood P, Levi AD. Safety of Autologous Human Schwann Cell Transplantation in Subacute Thoracic Spinal Cord Injury. J Neurotrauma. 2017 Nov 1;34(21):2950-2963. doi: 10.1089/neu.2016.4895. Epub 2017 Mar 21. PMID 28225648
- See also: Related Info — http://www.themiamiproject.org